CLINICAL TRIAL: NCT06735625
Title: Pilot Study "AHSP as a Biomarker of Sickle Cell Disease in a Population of Adults and Children"
Acronym: AHSPDREP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier de Saint-Denis (Other)
Collaborators: Inserm U955 (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 0048_MEDECINE INTERNE_PEDIATRI; 2023-A02784-41 (Registry Identifier: IDRCB)
Record Dates: First submitted 2024-12-11; First posted 2024-12-16 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2024-07

CONDITIONS: in Relation to Sickle Cell Disease
Keywords: AHSP; Sickle Cell Disease; SS Phenotype; Sβ0 Phenotype
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Intervention Model Description: 30 sickle cell patients over 15 and a half years old with SS or Sβ0 phenotype 30 control patients over 15 and a half years old without hemoglobin abnormalities, recruited at the hospital 20 pediatric sickle cell patients (aged between 3 and 15 and a half years) with SS or Sβ0 phenotype 20 pediatric control patients (aged between 3 and 15 and a half years) without hemoglobin abnormalities, recruited at the hospital
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- sickle cell patients over 15 and a half years old (Experimental): sickle cell patients over 15 and a half years old with SS or Sβ0 phenotype
  Interventions: Biological: Measurement of AHSP concentration
- control patients over 15 and a half years old (Other): control patients over 15 and a half years old without hemoglobin abnormalities, recruited at the hospital
  Interventions: Biological: Measurement of AHSP concentration
- pediatric sickle cell patients (aged between 3 and 15 and a half years) (Experimental): pediatric sickle cell patients (aged between 3 and 15 and a half years) with SS or Sβ0 phenotype
  Interventions: Biological: Measurement of AHSP concentration
- pediatric control patients (aged between 3 and 15 and a half years) (Other): pediatric control patients (aged between 3 and 15 and a half years) without hemoglobin abnormalities, recruited at the hospital
  Interventions: Biological: Measurement of AHSP concentration

INTERVENTIONS:
Biological: Measurement of AHSP concentration — Pseudonymization and identification of research samples EDTA tube of 4 mL for patients over 15 and a half years old, and 2 EDTA tubes of 2 mL for children aged 3 to 15 and a half years, totaling 4 mL) by Team 4 according to the procedure in force at the URC.
  The 4 mL research sample will then be divided into 1 mL fractions by a technician in the laboratory and stored at -80°C in the medical biology laboratory.

SUMMARY:
Evaluation of AHSP concentration in total blood as a biomarker in adult and pediatric sickle cell patients

DETAILED DESCRIPTION:
Research involving non-interventional humans. Selection and inclusion of patients by CHSD investigators. Collection of clinical data by investigators and CHSD URC staff.

Biochemical and hematological measurements by the CHSD medical biology laboratory for "care" samples Pseudonymization of 4 mL "research" samples by the URC then fractionation of the samples by 1 mL, and storage at -80°C within the medical biology laboratory of the CHSD.

Transport of samples at -80°C to team 1 of Dr Baudin-Creuza (Créteil). Preparation of genomic DNA from a 1 mL fraction then α and β globin genotyping by Dr Pissard.

Measurement of the AHSP concentration from the other fractions. Comparison of the AHSP concentration according to the group of subjects, and with the different parameters, then correlation analysis

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for Sickle Cell Patients

1. Adults: > 15 years and 6 months
2. Pediatrics: ≥ 3 years and ≤ 15 years and 6 months
3. Known SS or Sβ0 phenotypes

Inclusion Criteria for Control Patients.

1 -Adults: > 15 years and 6 months /Pediatrics: ≥ 3 years and ≤ 15 years and 6 months 2-Absence of Hemoglobinopathy 3-Follow-up for one of the following conditions (adults): Evaluation of hematological disease excluding hemoglobinopathy, evaluation of prolonged fever or inflammatory syndrome, initial or episodic evaluation of an auto-inflammatory disease or systemic disease, general health deterioration

-Follow-up for one of the following conditions (pediatrics): Suspected precocious puberty, growth delay, or neurodevelopmental disorder

4-Blood sample planned as part of medical care

Exclusion Criteria:

1. Hemoglobin disorder other than sickle cell disease (Criteria for Sickle Cell Patients)
2. Hemoglobinopathies other than sickle cell disease (Criteria for Control Patients)
3. Transfusion less than 3 months ago
4. Chronic active viral disease: hepatitis B, C, HIV
5. Current infections or known inflammatory pathologies
6. Known hyper or hypothyroidism or subject treated with levothyroxine
7. Active tumor pathology or remission for less than 5 years
8. Oral corticosteroid therapy in progress
9. Participation in interventional biomedical research
10. Opposition to participation in research by the patient if he is an adult, or by one of the two parents if the patient is a minor.
11. Non-affiliation to a social security system

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-03-06 (Actual); Primary Completion 2026-03-20 (Estimated); Study Completion 2027-01-20 (Estimated)

PRIMARY OUTCOMES:
AHSP concentrations measured in patients | 6 MONTH
  Comparison of AHSP concentrations measured in total blood between:
  Those of adult sickle cell patients and those of adult control patients without sickle cell disease Those of pediatric sickle cell patients and those of pediatric control patients without sickle cell disease

SECONDARY OUTCOMES:
Correlation analysis | 6 MONTH
  Correlation analysis between the AHSP parameter and the clinical-biological, therapeutic, and genetic parameters of adult and pediatric sickle cell patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier de Saint-Denis, Saint-Denis, France

REFERENCES:
- See also: Decreased sickle red blood cell adhesion to laminin by hydroxyurea is associated with inhibition of Lu/BCAM protein phosphorylation — https://pubmed.ncbi.nlm.nih.gov/20566895/
- See also: F. Clinical management of adult sickle-cell disease. Curr Opin Hematol — https://pubmed.ncbi.nlm.nih.gov/22357165/
- See also: 2D DIGE based proteomics study of erythrocyte cytosol in sickle cell disease: altered proteostasis and oxidative stress — https://pubmed.ncbi.nlm.nih.gov/24030922/
- See also: Alpha-hemoglobin stabilizing protein (AHSP), a kinetic scheme of the action of a human mutant, AHSPV56G — https://pubmed.ncbi.nlm.nih.gov/20371604/